CLINICAL TRIAL: NCT05205395
Title: Relationship Between Q-tip Test and Urethral Hypermobility on Perineal Ultrasound for Women With Urodynamic Stress Incontinence
Brief Title: Relationship Between Q-tip Test and Urethral Hypermobility
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(I)20210275
Record Dates: First submitted 2021-12-21; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Urodynamic Stress Incontinence
Keywords: Urodynamic stress incontinence; Q-tip test; Transperineal ultrasound; Urethral hypermobility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with stress incontinence: Women with urodynamic stress incontinence (USI) scheduled for mid-urethral sling surgery in the urogynecological department of a tertiary referral center were recruited.
  Interventions: Diagnostic Test: Transperineal ultrasound

INTERVENTIONS:
Diagnostic Test: Transperineal ultrasound — Ultrasonography was used with curved linear-array transducer placed between the major labia and underneath the external urethral orifice. The measurement was done on the midsagittal plane to obtain the image of pubic symphysis, urethra, and bladder in a view. Ultrasonic measurement of the overall rest-stress distance was define as the linear distance of bladder neck position change from resting status to maximal strain.

SUMMARY:
Q-tip test was applied for evaluation of urethral hypermobility (UH) in stress-incontinent women. It is still unknown whether there is an alternative method for the assessment of UH in a less invasive way or not.

We aim to assess the correlation between the overall rest-stress distance measured by transperineal ultrasound (TPUS) and Q-tip test angle in women with urodynamic stress incontinence (USI) scheduled for mid-urethral sling surgery (MUS), and determine a cut off value of rest-stress distance for predicting UH.

DETAILED DESCRIPTION:
Between January 2009 and January 2014, women with urodynamic stress incontinence (USI) scheduled for mid-urethral sling surgery in the urogynecological department of a tertiary referral center were recruited. A retrospective chart review was performed. This study received approval from the Institutional Review Board of Kaohsiung Medical University Hospital (ID:KMUHIRB-E(I)-20210275), by which relevant guidelines and regulations were followed accordingly. Informed consent was obtained from all participants before surgeries. The Q-tip test was performed via a cotton swab with the patient in a 45-degree reclining. After lubricated with 2% lidocaine jelly, the cotton swab was inserted with the tip over bladder neck. The angle changes from rest to maximal straining were obtained for 3 times, and the maximum of angle change was recorded. The TPUS was performed by two experienced urogynecologist according to KMUH-TPUS protocol. The Voluson General Electric Sonography, expert 730 type (GE, Healthcare Ultrasound, Zipf, Austria) Ultrasonography was used with 3.5 MHZ curved linear-array transducer placed between the major labia and underneath the external urethral orifice. The measurement was done on the midsagittal plane to obtain the image of pubic symphysis, urethra, and bladder in a view. Ultrasonic measurement of the overall rest-stress distance was define as the linear distance of bladder neck position change from resting status to maximal strain. The rest-stress distance was obtained for 3 times, and the maximum of distance was recorded. The primary outcome of this study was the correlation between the angle of Q-tip test and the overall rest-stress distance of bladder neck in TPUS. The secondary outcome was the optimal cut off value of the rest-stress distance to predict UH.

ELIGIBILITY:
Inclusion Criteria:

* Women with urodynamic stress incontinence (USI)
* Scheduled for mid-urethral sling surgery

Exclusion Criteria:

* Women with more or equal to stage 2 pelvic organ prolapse (POP) defined by POP-quantification system (POP-Q) and received concomitant transvaginal mesh (TVM) surgery
* Women with incomplete ultrasound records

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2009 and January 2014, a total of 258 women with urodynamic stress incontinence (USI) scheduled for mid-urethral sling surgery in the urogynecological department of a tertiary referral center were recruited. A retrospective chart review was performed. Women with more or equal to stage 2 pelvic organ prolapse (POP) defined by POP-quantification system (POP-Q) and received concomitant transvaginal mesh (TVM) surgery were excluded. Women with incomplete ultrasound records were also excluded.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
Q-tip test and therest-stress distance | January 2009 to January 2014
  The correlation between the angle of Q-tip test and the overall rest-stress distance of bladder neck

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yu Long, Principal Investigator — Kaohsiung Municipal Siaogang Hospital

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Result] Nygaard IE, Heit M. Stress urinary incontinence. Obstet Gynecol. 2004 Sep;104(3):607-20. doi: 10.1097/01.AOG.0000137874.84862.94. PMID 15339776
- [Result] DeLancey JO. Structural support of the urethra as it relates to stress urinary incontinence: the hammock hypothesis. Am J Obstet Gynecol. 1994 Jun;170(6):1713-20; discussion 1720-3. doi: 10.1016/s0002-9378(94)70346-9. PMID 8203431
- [Result] Crystle CD, Charme LS, Copeland WE. Q-tip test in stress urinary incontinence. Obstet Gynecol. 1971 Aug;38(2):313-5. No abstract available. PMID 5105346
- [Result] Dietz HP. Pelvic floor ultrasound: a review. Am J Obstet Gynecol. 2010 Apr;202(4):321-34. doi: 10.1016/j.ajog.2009.08.018. PMID 20350640
- [Result] Walters MD, Shields LE. The diagnostic value of history, physical examination, and the Q-tip cotton swab test in women with urinary incontinence. Am J Obstet Gynecol. 1988 Jul;159(1):145-9. doi: 10.1016/0002-9378(88)90510-8. PMID 3394734
- [Result] Yun JH, Kim JH, Park S, Lee C. Changes in the Q-tip angle in relation to the patient position and bladder filling. BMC Urol. 2015 Oct 7;15:101. doi: 10.1186/s12894-015-0096-4. PMID 26446765
- [Result] Chen GD, Su TH, Lin LY. Applicability of perineal sonography in anatomical evaluation of bladder neck in women with and without genuine stress incontinence. J Clin Ultrasound. 1997 May;25(4):189-94. doi: 10.1002/(sici)1097-0096(199705)25:43.0.co;2-a. PMID 9142618
- [Result] Lin KL, Juan YS, Lo TS, Liu CM, Tsai EM, Long CY. Three-dimensional ultrasonographic assessment of compression effect on urethra following tension-free vaginal tape and transobturator tape procedures. Ultrasound Obstet Gynecol. 2012 Apr;39(4):452-7. doi: 10.1002/uog.9071. PMID 21656867